CLINICAL TRIAL: NCT00346073
Title: A Study to Evaluate Immunogenicity and Safety of Boostrix Compared to Adacel When Administered as a Booster Vaccination in Adults Aged 19 to 64 Years of Age
Brief Title: Safety and Immunogenicity of GSK's Tdap Vaccine (Boostrix) in Adults Aged 19 to 64 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 106316
Record Dates: First submitted 2006-06-28; First posted 2006-06-29 (Estimated); Results first posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-02

CONDITIONS: Acellular Pertussis; Diphtheria; Tetanus
Keywords: Prophylaxis for diphtheria, tetanus, pertussis; Immunogenicity, booster, dTpa
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough | interventions — Boostrix; adacel

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Boostrix Group (Experimental): Subjects, male or female, between, and including, 19 and 64 years of age received a single dose of Boostrix® vaccine administered intramuscularly in the deltoid region of the non-dominant upper arm at Day 0.
  Interventions: Biological: Boostrix™
- Adacel Group (Experimental): Subjects, male or female, between, and including, 19 and 64 years of age received a single dose of Adacel™ vaccine administered intramuscularly in the deltoid region of the non-dominant upper arm at Day 0.
  Interventions: Biological: ADACEL®

INTERVENTIONS:
Biological: Boostrix™ — Combined Reduced Antigen Content Diphtheria, Tetanus, Acellular Pertussis Vaccine
  Arms: Boostrix Group
Biological: ADACEL® — Sanofi Pasteur
  Arms: Adacel Group

SUMMARY:
GSK Biologicals' dTpa vaccine has recently been approved by the US Food and Drug Administration (FDA) for booster vaccination of adolescents aged 10 to 18 years. The ACIP has recently issued provisional recommendations for universal adult Tdap vaccination. The current study will provide pivotal data in support of extending the age range for Boostrix vaccine to include adults 19-64 years of age.

ELIGIBILITY:
Inclusion Criteria:

* A healthy male or female, 19 to 64 years of age (not having reached the 65th birthday) at the time of study vaccination.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding administration of study vaccine, or planned use during the active phase of the study.
* Chronic administration of immunosuppressants or within six months prior to administration of study vaccine.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within 30 days of administration of study vaccine (with the exception of an influenza vaccine).
* Administration of a diphtheria-tetanus (Td) booster within previous five years.
* Administration of Tdap vaccine at any time prior to study entry. History of serious allergic reaction (e.g. anaphylaxis) following any other tetanus toxoid, diphtheria toxoid or pertussis-containing vaccine or any component of the study vaccines.

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2337 (Actual)
Dates: Start 2006-07-13 (Actual); Primary Completion 2007-03-01 (Actual); Study Completion 2007-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (39):
- United States (39):
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Peoria, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tempe, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Pueblo, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Boise, Idaho
  - GSK Investigational Site, Peoria, Illinois
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Richland, Michigan
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Alliance, Nebraska
  - GSK Investigational Site, North Platte, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Bismarck, North Dakota
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Grove City, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, West Jordan, Utah
  - GSK Investigational Site, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Blatter M, Friedland LR, Weston WM, Li P, Howe B. Immunogenicity and safety of a tetanus toxoid, reduced diphtheria toxoid and three-component acellular pertussis vaccine in adults 19-64 years of age. Vaccine. 2009 Jan 29;27(5):765-72. doi: 10.1016/j.vaccine.2008.11.028. Epub 2008 Nov 27. PMID 19041352
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 106316 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 106316 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 106316 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 106316 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 106316 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 106316 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 2337 subjects were enrolled into the study. Of these, 53 subjects were allocated subject numbers, but did not receive study vaccination.
Period: Overall Study
Arm/Group | Boostrix Group | Adacel Group
Started | 1522 | 762
Completed | 1481 | 738
Not Completed | 41 | 24
Not completed — Serious Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 39 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Boostrix Group | Adacel Group | Total
Number analyzed (Participants) | 1522 | 762 | 2284
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.9 (13.64) | 40.1 (13.51) | 39.97 (13.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 946 | 479 | 1425
  Male | 576 | 283 | 859
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: African heritage/African American | 126 | 61 | 187
  Geographic ancestry: American Indian or Alaskan native | 6 | 5 | 11
  Geographic ancestry: Asian - Central/South Asian heritage | 1 | 0 | 1
  Geographic ancestry: Asian - East Asian heritage | 2 | 1 | 3
  Geographic ancestry: Asian - Japanese heritage | 3 | 0 | 3
  Geographic ancestry: Asian - South East Asian heritage | 6 | 3 | 9
  Geographic ancestry: Native Hawaiian or other Pacific islander | 6 | 3 | 9
  Geographic ancestry: White - Arabic/North African heritage | 19 | 13 | 32
  Geographic ancestry: White - Caucasian/European heritage | 1281 | 635 | 1916
  Geographic ancestry: Not specified | 72 | 41 | 113

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroprotected Subjects With Anti-diphteria (Anti-D) and Anti-tetanus (Anti-T) Antibodies
Description: A seroprotected subject is defined as a vaccinated subject with anti-D and anti-T antibody concentration greater than or equal to ( ≥) 0.1 international units per milliliter (IU/mL).
Time Frame: At Month 1
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects who met all eligibility criteria, who complied with the protocol requirements and for whom immunogenicity measures were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group
Number analyzed (Participants) | 1445 | 728
Participants
  Anti-D: number analyzed (Participants) | 1444 | 727
  Anti-D | 1418 | 717
  Anti-T | 1439 | 728
Statistical Analysis 1: Comparison: Boostrix Group vs Adacel Group; The non-inferiority of Boostrix® vaccine compared to Adacel™ vaccine, with respect to the percentage of subjects with anti-diphtheria (anti-D) antibody concentrations greater than or equal to (≥) 0.1 IU/mL, one month after vaccination; Test type: Non-Inferiority — The primary objective of non-inferiority was met if the lower limit of the 95% confidence intervals (CIs), between the two groups (Boostrix Group - Adacel Group) were greater than or equal to (≥) -10%; Difference in percentage = -0.43, 95% CI 2-sided [-1.47 to 0.84]
Statistical Analysis 2: Comparison: Boostrix Group vs Adacel Group; The non-inferiority of Boostrix® vaccine compared to Adacel™ vaccine, with respect to the percentage of subjects with anti-tetanus (anti-T) antibody concentrations greater than or equal to (≥) 0.1 IU/mL, one month after vaccination; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in percentage = -0.42, 95% CI 2-sided [-0.9 to 0.11]

2. Primary Outcome: Number of Seropositive Subjects With Anti-tetanus (Anti-T) Antibodies
Description: A seropositive subject was a subject whose antibody concentration was greater than or equal to the cut-off value. Cut-off values assessed were greater than or equal to 1.0 international units per milliliter (IU/mL).
Time Frame: At Month 1
Population: The analysis was performed on the According-To-Protocol cohort for immunogenicity, which included all evaluable subjects who met all eligibility criteria, who complied with the protocol requirements and for whom immunogenicity measures were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group
Number analyzed (Participants) | 1445 | 728
Participants | 1420 | 723
Statistical Analysis 1: Comparison: Boostrix Group vs Adacel Group; The non-inferiority of Boostrix® vaccine compared to Adacel™ vaccine, with respect to the percentage of subjects with anti-tetanus (anti-T) antibody concentrations greater than or equal to (≥) 1.0 IU/mL, one month after vaccination; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in percentage = -1.04, 95% CI 2-sided [-1.97 to 0]

3. Primary Outcome: Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Hemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN) Antibody Concentrations
Description: Concentrations are presented as geometric mean concentrations (GMCs) and expressed in enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: At Month 1
Population: The analysis was performed on the According-To-Protocol cohort for immunogenicity, which included all evaluable subjects who met all eligibility criteria, who complied with the protocol requirements and for whom immunogenicity measures were available. The primary outcome results only refer to subjects who received a Boostrix vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Boostrix Group | Adacel Group
Number analyzed (Participants) | 1444 | 726
EL.U/mL
  Anti-PT: number analyzed (Participants) | 1431 | 722
  Anti-PT | 63.6 [60.1 to 67.4] | 32.2 [29.6 to 35.1]
  Anti-FHA: number analyzed (Participants) | 1443 | 724
  Anti-FHA | 624.4 [593.9 to 656.6] | 368.4 [344.3 to 394.2]
  Anti-PRN | 401.0 [368.5 to 436.3] | 351.9 [315.7 to 392.2]

4. Primary Outcome: Number of Subjects With Booster Responses for Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Hemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN) Antibodies
Description: Booster responses for anti-PT, anti-FHA and anti-PRN antibodies were defined as: for initially seronegative subjects (pre-vaccination concentration below cut-off: smaller than (<) 5 EU/mL): antibody concentrations at least four times the cut-off (post-vaccination concentration greater than or equal to (≥) 20 EU/mL), one month after vaccination; for initially seropositive subjects with pre-vaccination concentration ≥ 5 EU/mL and < 20 EU/mL: an increase in antibody concentrations of at least four times the pre-vaccination concentration one month after vaccination; and for initially seropositive subjects with pre-vaccination concentration ≥ 20 EU/mL: an increase in antibody concentrations of at least two times the pre-vaccination concentration, one month after vaccination.
Time Frame: At Month 1
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group
Number analyzed (Participants) | 1441 | 725
Participants
  Anti-PT: number analyzed (Participants) | 1419 | 717
  Anti-PT | 1095 | 338
  Anti-FHA: number analyzed (Participants) | 1433 | 714
  Anti-FHA | 1388 | 671
  Anti-PRN | 1343 | 665
Statistical Analysis 1: Comparison: Boostrix Group; Demonstration that anti-PT booster response occurred in at least 80% of adults receiving a single dose of Boostrix® vaccine, one month after vaccination. Criterion for evaluation: one month after vaccination, the lower limit of the 95% confidence interval (CI) for the percentage of subjects with a booster response was greater than or equal to (≥) 80%; Test type: Superiority; Booster response = 77.2, 95% CI 2-sided [74.9 to 79.3]
Statistical Analysis 2: Comparison: Boostrix Group; Demonstration that anti-FHA booster response occurred in at least 80% of adults receiving a single dose of Boostrix® vaccine, one month after vaccination. Criterion for evaluation: one month after vaccination, the lower limit of the 95% confidence interval (CI) for the percentage of subjects with a booster response was greater than or equal to (≥) 80%; Test type: Superiority; Booster response = 96.9, 95% CI 2-sided [95.8 to 97.7]
Statistical Analysis 3: Comparison: Boostrix Group; Demonstration that anti-PRN booster response occurred in at least 80% of adults receiving a single dose of Boostrix® vaccine, one month after vaccination. Criterion for evaluation: one month after vaccination, the lower limit of the 95% confidence interval (CI) for the percentage of subjects with a booster response was greater than or equal to (≥) 80%; Test type: Superiority; Booster response = 93.2, 95% CI 2-sided [91.8 to 94.4]

5. Secondary Outcome: Number of Seropositive Subjects With Anti-diphteria (Anti-D) Antibodies
Description: A seropositive subject was a subject whose antibody concentration was greater than or equal to the cut-off value. Cut-off values assessed were greater than or equal to (≥) 1.0 international units per milliliter (IU/mL).
Time Frame: At Month 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group
Number analyzed (Participants) | 1444 | 727
Participants | 1269 | 669

6. Secondary Outcome: Number of Subjects With Booster Responses for Anti-diphteria (Anti-D) and Anti-tetanus (Anti-T)
Description: Booster responses for anti-D and anti-T antibodies were defined as: for initially seronegative subjects (pre-vaccination concentration below cut-off: smaller than (<) 0.1 IU/mL): antibody concentrations at least four times the cut-off (post-vaccination concentration greater than or equal to (≥ 0.4 IU/mL), one month after vaccination; and for initially seropositive subjects (pre-vaccination concentration ≥ 0.1 IU/mL): an increase in antibody concentrations of at least four times the pre-vaccination concentration one month after vaccination.
Time Frame: At Month 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group
Number analyzed (Participants) | 1444 | 727
Participants
  Anti-D: number analyzed (Participants) | 1438 | 720
  Anti-D | 1116 | 566
  Anti-T | 704 | 441

7. Secondary Outcome: Anti-diphteria (Anti-D) and Anti-tetanus (Anti-T) Antibody Concentrations
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: At Month 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Boostrix Group | Adacel Group
Number analyzed (Participants) | 1445 | 728
EL.U/mL
  Anti-D: number analyzed (Participants) | 1444 | 727
  Anti-D | 4.7 [4.4 to 5.1] | 5.0 [4.6 to 5.4]
  Anti-T | 8.5 [8.1 to 8.9] | 13.3 [12.5 to 14.1]

8. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 50 millimeters (mm) of injection site.
Time Frame: During the 15-day period (Day 0-14) following vaccination
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects with at least one vaccine administration documented and with the symptom sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group
Number analyzed (Participants) | 1480 | 741
Participants
  Pain, Any | 903 | 513
  Pain, Grade 3 | 24 | 17
  Redness, Any | 313 | 201
  Redness, ≥ 50 mm | 23 | 17
  Swelling, Any | 260 | 190
  Swelling, ≥ 50 mm | 21 | 21

9. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, fever [defined as temperature measured orally, greater than or equal to (≥) 37.5 degrees Celsius (°C)], gastrointestinal symptoms [gastro sympt.] and headache. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 15-day period (Day 0-14) following vaccination
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group
Number analyzed (Participants) | 1480 | 741
Participants
  Fatigue, Any | 416 | 214
  Fatigue, Grade 3 | 37 | 9
  Fatigue, Related | 251 | 151
  Fever (orally), ≥37.5 °C | 82 | 59
  Fever (orally), ≥39 °C | 1 | 3
  Fever, Related | 40 | 28
  Gastro sympt., Any | 235 | 130
  Gastro sympt., Grade 3 | 18 | 10
  Gastro sympt., Related | 125 | 67
  Headache, Any | 445 | 230
  Headache, Grade 3 | 32 | 11
  Headache, Related | 245 | 143

10. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day period (Days 0-30) following vaccination
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group
Number analyzed (Participants) | 1522 | 762
Participants | 271 | 169

11. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs).
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the active phase of the study (Day 0 - Day 30)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group
Number analyzed (Participants) | 1522 | 762
Participants | 9 | 2

12. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 11
Time Frame: During the extended safety follow-up (ESFU) phase (Day 31 - Month 6)
Population: The analysis was performed on the Extended Safety Follow Up (ESFU) cohort, which included all the subjects for whom the ESFU contact was completed. Two subjects were not contacted after the active phase of study, but had SAEs reported in the ESFU period.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group
Number analyzed (Participants) | 1445 | 719
Participants | 12 | 11

13. Secondary Outcome: Number of Subjects Reporting Hospitalizations
Description: Hospitalization signified that the subject had been detained (usually involving at least an overnight stay) at the hospital or emergency ward for observation and/or treatment that would not have been appropriate in the physician's office or out patient setting.
Time Frame: During the extended safety follow-up (ESFU) period (from Day 31 to Month 6)
Population: The analysis was performed on the Extended Safety Follow Up (ESFU) cohort, which included all the subjects for whom the ESFU contact was completed.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group
Number analyzed (Participants) | 1444 | 718
Participants | 13 | 10

14. Secondary Outcome: Number of Subjects Reporting Emergency Room Visits
Description: Emergency room visits refer to AEs requiring immediate medical attention.
Time Frame: During the extended safety follow-up (ESFU) period (from Day 31 to Month 6)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group
Number analyzed (Participants) | 1444 | 718
Participants | 13 | 6

15. Secondary Outcome: Number of Subjects Reporting the Onset of New Chronic Illnesses
Description: New onset chronic illnesses include diabetes, asthma, allergies, autoimmune diseases.
Time Frame: During the extended safety follow-up (ESFU) period (from Day 31 to Month 6)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group
Number analyzed (Participants) | 1444 | 718
Participants | 2 | 3

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 15-day (Day 0-14) follow-up period after vaccination; Unsolicited AEs: during the 31-day (Day 0-30) follow-up period after vaccination; SAEs: during the entire study period, including the ESFU phase (Month 0 - Month 6).
Arm/Group | Boostrix Group | Adacel Group
All-Cause Mortality (participants affected / at risk) | 1/1522 | 1/762
Serious Adverse Events (participants affected / at risk) | 21/1522 | 13/762
Other Adverse Events (participants affected / at risk) | 1108/1522 | 595/762
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Boostrix Group (N=1522) | Adacel Group (N=762)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Schizoaffective disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Menometrorrhagia (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Herpes oesophagitis (Infections and infestations) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Localized infection (Infections and infestations) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Meningitis aseptic (Infections and infestations) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin graft (Surgical and medical procedures) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urge incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Boostrix Group (N=1522) | Adacel Group (N=762)
Erythema (Skin and subcutaneous tissue disorders) | 313 (313) | 201 (201)
Fatigue (General disorders) | 419 (420) | 214 (214)
Gastrointestinal disorder (Gastrointestinal disorders) | 235 (235) | 130 (130)
Headache (Nervous system disorders) | 448 (450) | 230 (232)
Pain (General disorders) | 905 (917) | 516 (530)
Pyrexia (General disorders) | 82 (82) | 60 (61)
Swelling (General disorders) | 261 (261) | 190 (191)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.